CLINICAL TRIAL: NCT04051749
Title: Incidence, Predictors and Validation of Risk Scores to Predict Myocardial Infarction After Noncardiac Vascular Surgery, a Cohort Prospective Study
Brief Title: Incidence, Predictors and Validation of Risk Scores to Predict Myocardial Infarction After Noncardiac Vascular Surgery
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Pedro Reis, Principal Investigator, Centro Hospitalar De São João, E.P.E.
Other Study IDs: CES 04-15
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Complication of Surgical or Medical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients submitted to VS
  Interventions: Procedure: Noncardiac Vascular Surgery

INTERVENTIONS:
Procedure: Noncardiac Vascular Surgery — Noncardiac Vascular Surgery

SUMMARY:
Evaluate the incidence and predictors of post-operative mortality after noncardiac Vascular Surgery and compare the performance of existing risk scores.

ELIGIBILITY:
Inclusion Criteria:

* Elective arterial Vascular Surgery
* Patients > 18 years

Exclusion Criteria:

* Urgent/Emergent Surgery
* Patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients submitted to elective arterial VS
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Major Cardiac Events | 30-day

SECONDARY OUTCOMES:
Mortality | 30-day

REFERENCES:
- [Derived] Reis P, Mourao J, Abelha F. Reply to the commentary on "Incidence, predictors and validation of risk scores to predict postoperative mortality after noncardiac vascular surgery, a prospective cohort study" [Int. J. Surg. 77 (2020) 181-2]. Int J Surg. 2020 Jul;79:47-49. doi: 10.1016/j.ijsu.2020.04.072. Epub 2020 May 11. No abstract available. PMID 32438070